CLINICAL TRIAL: NCT03560271
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 2 Study to Evaluate the Efficacy and Safety of Cyclo-Z in Subjects With Type 2 Diabetes
Brief Title: A Phase 2 Study of Cyclo-Z in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovMetaPharma Co., Ltd. (Industry)
Collaborators: InClin, Inc. (Unknown); FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMP-CYZ-P2-002
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Z 008; somatostatin, cyclic hexapeptide(Phe-Phe-Trp-Lys-Thr-Phe)-; Zinc

STUDY DESIGN:
Intervention Model Description: Subject will be assigned to either 6 mg Cyclo-Z, 15 mg Cyclo-Z or placebo for the duration of study treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, sponsor, and subject will be blinded to study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose A (Experimental): Cyclo-Z containing 23 mg zinc plus 6 mg CHP
  Interventions: Drug: Cyclo-Z
- Dose B (Experimental): Cyclo-Z containing 23 mg zinc plus 15 mg CHP
  Interventions: Drug: Cyclo-Z
- Dose C (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cyclo-Z — Cyclo (His-Pro) and zinc
  Other Names: CHP plus zinc
  Arms: Dose A; Dose B
Other: Placebo — Matching placebo
  Arms: Dose C

SUMMARY:
This is a double-blind, randomized, placebo-controlled, parallel-group comparison study to evaluate the efficacy and safety of Cyclo-Z vs. placebo in adult subjects with type 2 diabetes. Approximately 20 clinical sites may be utilized in the United States so that approximately 300 subjects (a potential 20% screening failure rate) may be screened for total 28-week study period (2 weeks for screening, 24 weeks for treatment, and 2 weeks for safety follow-up).

DETAILED DESCRIPTION:
Insulin degrading enzyme (IDE) is a zinc-containing enzyme that regulates degradation of internalized insulin and the maintenance of insulin sensitivity. Diabetic animals and humans are zinc deficient due to impaired intestinal zinc absorption and hyperzincuria. If endosomal IDE levels are inadequate, undigested insulin will remain in the cytosol and prevent insulin signal transduction. Cyclo-Z enhances IDE synthesis and stimulates insulin degradation. Although Cyclo (his-pro) (CHP) or zinc alone are somewhat effective in the control of blood glucose metabolism, based on the available literature and previous background studies, it is hypothesized that the combination of CHP and zinc in Cyclo-Z work synergistically to ameliorate insulin resistance in diabetic and obese subjects mainly by stimulating IDE synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 or older.
* Subjects diagnosed with type 2 diabetes mellitus (DM) according to the American Diabetes Association (ADA) criteria.
* Subjects treated with stable doses of insulin and/or other hypoglycemic agent(s) for type 2 diabetes mellitus for at least 2 months prior to randomization and who agree to stay on stable doses of anti-diabetes agents during the study.
* Subjects whose fasting blood glucose levels are reasonably stable for at least 2 months prior to randomization and during the 2-week screening period.
* Subjects who have Hemoglobin A1c levels of 7.5 to 10.0 % at Screening and a fasting plasma glucose less than 310 mg/dL.
* Subjects who can give written informed consent.
* Subjects who are willing and able to monitor their blood glucose concentrations with a home glucose monitor (before breakfast and 2 hours after dinner).
* Female subjects must be either:

  * Surgically sterile (i.e., have had bilateral tubal ligation, hysterectomy, or bilateral oophorectomy) at least 6 months before randomization, or
  * Post-menopausal for at least 12 months prior to Screening, or
  * If of childbearing potential and sexually active, must agree to use adequate contraception from Screening to completion of the study.

Exclusion Criteria:

* Subjects who have any significant DM-related end-organ damages.
* Subjects who have a history of diabetic ketoacidosis or hyperosmolar non-ketotic coma.
* Subjects who have any disease likely to limit life span and/or increase risks of interventions such as:

  * Carotid B-mode ultrasound test results indicating clinically significant stenosis in the common carotid arteries requiring intervention by angioplasty or resection.
  * Cancer treatment in the past 5 years, with the exception of cancers which have been cured, and carry a good prognosis.
  * Infectious disease: HIV positivity, active tuberculosis, or pneumonia.
* Subjects with evidence of clinically significant cardiovascular or cerebrovascular disease, including (but not limited to):

  * Hospitalization for the treatment of heart disease in the past 12 months.
  * New York Heart Association Functional Class > 2.
  * Left bundle branch block on ECG at Screening.
  * Third degree atrioventricular block on ECG at Screening.
  * Stroke or transient ischemic attack in the past 12 months.
* Subjects with uncontrolled hypertension with average systolic blood pressure of ≥ 160 mmHg or diastolic blood pressure ≥ 95 mmHg at Screening and Baseline.
* Subjects with pulse rate ≥ 95 beats per minute at Screening and Baseline.
* Subjects who have or had any of the following conditions related to gastrointestinal disease:

  * Chronic hepatitis or cirrhosis.
  * Episode of alcoholic hepatitis or pancreatitis.
  * Inflammatory bowel disease or irritable bowel syndrome.
  * Significant abdominal surgery (e.g., gastrectomy, gastric bypass) in the past 2 months.
* Serum creatinine ≥ 1.5 mg/dL for males or ≥ 1.4 mg/dL for females.
* Hemoglobin ≤ 12 g/dL for males or ≤ 10 g/dL for females.
* Subjects who have chronic obstructive airway disease or asthma requiring daily inhaled corticosteroid therapy or home use oxygen.
* Subjects who have any of the following conditions or behaviors likely to affect the conduct of the study:

  * Weight loss of > 10% in the past 6 months.
  * Unable to walk without assisted device.
  * Major psychiatric disorder which would impede conduct of the research.
  * Excessive alcohol intake (i.e., more than 2 drinks/day).
  * Use of illicit drugs or drugs of abuse.
* Subjects who take any of the following medications:

  * Psychoactive agents such as monoamine oxidase inhibitors and antidepressants (e.g., lithium, Prozac, Zoloft, Serzone, Paxil, Effexor).
  * Any insulin sensitizers (thiazolidinediones - TZDs) such as Avandia, Actos or Duvie, etc.
* Subjects with any other clinically significant and/or unexplained abnormalities that, in the opinion of the Investigator, could impact the subject's ability to fully participate in or complete the study.
* Female subjects who have a positive serum pregnancy test at Screening, plan a pregnancy during study period, or are breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Glycosylated Hemoglobin (HbA1c) from Baseline at Week 24 | Day 1 to 24 weeks
  Change in HbA1c from Day 1 to Week 24

SECONDARY OUTCOMES:
Change from Baseline in HbA1c over time | Day 1 to 24 weeks
  Change in HbA1c over 24 weeks
Change from Baseline in fasting plasma glucose (FPG) levels over time | Day 1 to 24 weeks
  Change in FPG levels over 24 weeks
Change from Baseline in plasma insulin over time | Day 1 to 24 weeks
  Change in plasma insulin over 24 weeks
Proportion of subjects achieving HbA1c goal of < 7.0% at Week 24 | Day 1 to 24 weeks
  Percent of subjects who achieved HbA1c of <7% at Week 24
Proportion of subjects achieving HbA1c goal of < 6.5% at Week 24 | Day 1 to 24 weeks
  Percent of subjects who achieved HbA1c of <6.5% at Week 24
Proportion of subjects with decrease in HbA1c of ≥ 0.5% from Baseline at Week 24 | Day 1 to 24 weeks
  Percent of subjects who achieved HbA1c decrease at Week 24 of ≥ 0.5% from Day 1
Proportion of subjects with decrease in HbA1c of ≥ 1.0% from Baseline at Week 24 | Day 1 to 24 weeks
  Percent of subjects who achieved HbA1c decrease at Week 24 of ≥ 1.0% from Day 1

CONTACTS AND LOCATIONS:
Overall Officials: MiRa Huyghe, Study Director — NovMetaPharma Co., Ltd.
Locations (20):
- United States (20):
  - Study Site 29, Anniston, Alabama
  - Study Site 26, Birmingham, Alabama
  - Study Site 27, Chula Vista, California
  - Study Site 28, La Mesa, California
  - Study Site 10, Montclair, California
  - Study Site 23, North Hollywood, California
  - Study Site 13, Coral Gables, Florida
  - Study Site 19, DeLand, Florida
  - Study Site 14, Miami, Florida
  - Study Site 12, Miami Beach, Florida
  - Study Site 15, Orlando, Florida
  - Study Site 16, St. Petersburg, Florida
  - Study Site 21, Peachtree Corners, Georgia
  - Study Site 17, Snellville, Georgia
  - Study Site 20, North Dartmouth, Massachusetts
  - Study Site 30, Caro, Michigan
  - Study Site 24, Las Vegas, Nevada
  - Study Site 18, Cleveland, Ohio
  - Study Site 22, San Antonio, Texas
  - Study Site 11, San Antonio, Texas